CLINICAL TRIAL: NCT02349815
Title: Pharmacoepidemiological Study (Drug Utilization Study) of JAYDESS Use in Routine Clinical Practice in Sweden
Brief Title: JAYDESS Drug Utilization Study in Sweden
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 16903; JD1311SE (Other: Company internal)
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Contraception
Keywords: Drug Utilization Study
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Women prescribed JAYDESS in Sweden
  Interventions: Drug: Levonorgestrel (Jaydess, Skyla, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel (Jaydess, Skyla, BAY86-5028) — Women use Levonorgestrel (Jaydess, BAY86-5028) .

SUMMARY:
* To describe characteristics (demographic, clinical, social) of first time users of Jaydess
* To estimate the duration of use of Jaydess
* To study switching patterns, e.g. what are the hormonal contraceptive methods used before and what are the methods after discontinuing Jaydess
* To study off-label use of Jaydess

ELIGIBILITY:
Inclusion Criteria:

* Swedish women who were dispensed a JAYDESS from a Swedish Pharmacy anytime 2014-2017

Exclusion Criteria:

No exclusion criteria

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Duration of use of JAYDESS | Up to 6 years
Indication for use | At insertion

SECONDARY OUTCOMES:
Age at insertion and removal | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Sweden

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/